CLINICAL TRIAL: NCT00200668
Title: Comparison Between FDG-PET and MRI for the Assessment of Response to Intensive Chemotherapy in Multiple Myeloma Patients.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: BRD/04/6-H
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2008-06-09 (Estimated); Status verified 2008-06

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

INTERVENTIONS:
Drug: FDG = fluorodeoxyglucose

SUMMARY:
Comparison between FDG-PET and MRI for the assessment of response to intensive chemotherapy in multiple myeloma patients.

DETAILED DESCRIPTION:
First whole body FDG-PET scan and MRI before the start of the treatment. Second whole body FDG-PET scan and MRI after the end of the treatment. On a basis of patient, comparison between PET and MRI will be done tumoral site by site. Sensitivity, Specificity will be estimated for both techniques. In case of discrepancy, another imaging method or biopsy (if easy to perform) will be serve as standard of reference. Kappa coefficients and Mc Nemar test will be performed to compare the two methods. FDG = fluorodeoxyglucose FLUCIS® (Schering-CisBio® international)

ELIGIBILITY:
Inclusion Criteria:

* Patients from 18 to 65 years old.
* De novo histologically proven multiple myeloma.

Exclusion Criteria:

* No history of another cancer or of HIV
* No history of renal failure

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2005-03; Study Completion 2006-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Couturier, MD, Principal Investigator — Nantes University Hospital
Locations (1):
- Nantes University Hospital, Nantes, France